CLINICAL TRIAL: NCT07135752
Title: Comparison of Digital Biomarkers in Subjects With Radiologically Isolated Syndrome (RIS) and Multiple Sclerosis (MS) Patients With Clinically Normal Neurological Examination
Acronym: SPAM 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-PP-05
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Radiologically Isolated Syndromes; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple sclerosis (Other)
  Interventions: Other: Precision assessment
- Radiologically isolated syndrome (Other)
  Interventions: Other: Precision assessment

INTERVENTIONS:
Other: Precision assessment — Digital tools, imaging markers and biological markers

SUMMARY:
Radiologically Isolated Syndrome (RIS) is the preclinical stage of Multiple Sclerosis (MS). It is the incidental discovery of white matter abnormalities on brain or spinal cord magnetic resonance imaging (MRI), whose shape, topography and number are compatible with the radiological diagnostic criteria for MS. Individuals with a diagnosis of RIS should have a strictly normal neurological examination and, by definition, no history of clinical signs or symptoms that might suggest demyelinating disease. As recommended, patients with RIS benefit from brain and spinal cord MRI and a neurological examination by year to assess temporal dissemination (new T2 lesions and/or Gd+ lesions) and clinical manifestations. Epidemiological studies of RIS in the international RIS Consortium cohort have identified prognostic factors for conversion to multiple sclerosis. Five distinct long-term conversion risk factors were identified: age (subjects under 37 years of age at RIS diagnosis), the presence of oligoclonal bands (OCBs) on cerebrospinal fluid (CSF), the presence of infratentorial lesions, spinal cord lesions or gadolinium-enhanced lesions on index MRI. The presence of new T2 lesions on follow-up or contrast-enhanced MRI is also prognostic of progression to the clinical stage of the disease. The identification of other biomarkers at the preclinical stage of demyelinating disease should shed light on sensitive points in the transition from preclinical to clinical, relapsing-remitting or progressive multiple sclerosis. Studies have been realized to identify biological prognostic markers, but the availability of the assay technique remains limited to a small number of laboratories, and there is as yet no consensus on the practicalities of using this marker on an individual scale. The silent progression of MS, leading to irreversible disability in the absence of immunointervention, has now been demonstrated. The SPAM 1 study, a retrospective study based on data from the French MS Observatory (OFSEP) identified risk factors associated with the transition to secondary-progressive MS in RRMS patients treated early (within 5 years of diagnosis) with high-efficacy therapies. The SPAM 2 study evaluated imaging markers on a sample (100 patients) from the SPAM 1 study. Imaging techniques such as magnetic susceptibility sequences can be used to assess chronic demyelinating disease, but their availability in this field is limited to a small number of centers, and their reliability for use on an individual scale remains debatable. Following on from these 2 studies, the present SPAM 3 study aims to evaluate digital tools, imaging markers and biological markers for a better characterization of the disease and its prognosis in the early stages. Correlation studies on all biological, MRI and digital biomarkers have never been performed in the early stages of MS. There is therefore an unmet need for more relevant tools that can be more easily applied in everyday practice to monitor the evolution of the disease, both in its inflammatory and neurodegenerative expression, at the subclinical stage.

The investigators hypothesize that RIS patients and MS patients with normal neurological examination have similar results for the different biomarkers used in this study. If this hypothesis proves to be true, will it be necessary to wait for patients to present a specific, potentially disabling clinical event before offering them disease-modifying therapy in the context of pre-symptomatic MS?

ELIGIBILITY:
Inclusion Criteria:

RIS patients:

* Patients fulfilling the 2023 diagnostic RIS criteria
* Patients with a radiologically isolated syndrome (RIS) identified in local OFSEP databases (French Multiple Sclerosis Observatory)

MS patients:

- Patients with a normal neurological examination fulfilling the McDonald 2017 MS diagnostic criteria

For both groups:

- Patient affiliated to social security

Exclusion Criteria:

* The presence of motor, visual or cognitive deficits unrelated to MS that may interfere with test performance
* A diagnosis of progressive MS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparaison of digital biomarkers performance | 12 months
  To compare neurological performance based on precision assessment in a cohort of subjects with RIS compared with a group of MS patients with normal conventional neurological examination (EDSS=0).

SECONDARY OUTCOMES:
Comparaison of standard MRI biomarkers | Baseline and Month 12
  To compare in a cohort of subjects with RIS with a group of MS patients with normal conventional neurological examination (EDSS=0) the brain and cervical spinal cord imaging markers from standard MRI sequences: atrophy with white matter volume, gray matter volume and lesion volume at Baseline and Month 12
Comparaison of unconventional MRI biomarkers | Baseline and Month 12
  To compare in a cohort of subjects with RIS with a group of MS patients with normal conventional neurological examination (EDSS=0) the imaging markers from unconventional MRI sequences at baseline and at Month 12 : Central Vein Sign and paramagnetic RIM lesion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France